CLINICAL TRIAL: NCT00104299
Title: Rituximab Therapy for the Induction of Remission and Tolerance in ANCA-Associated Vasculitis (ITN021AI)
Brief Title: Rituximab for the Treatment of Wegener's Granulomatosis and Microscopic Polyangiitis
Acronym: RAVE
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Immune Tolerance Network (ITN) (Network); Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DAIT ITN021AI
Record Dates: First submitted 2005-02-24; First posted 2005-02-25 (Estimated); Results first posted 2011-08-25 (Estimated); Last update posted 2017-04-21 (Actual); Status verified 2017-03

CONDITIONS: Vasculitis; Wegener's Granulomatosis; Microscopic Polyangiitis
Keywords: ANCA; Vasculitis; Wegener's Granulomatosis; microscopic polyangiitis; ANCA-positive; ANCA-associated; ANCA-associated vasculitis; MPA
MeSH Terms: conditions — Vasculitis; Granulomatosis with Polyangiitis; Microscopic Polyangiitis; Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis | interventions — Rituximab; Cyclophosphamide; Control Groups; Azathioprine; Methylprednisolone; Prednisone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rituximab (Experimental)
  Interventions: Drug: Rituximab plus cyclophosphamide placebo (rituximab group); Drug: Methylprednisolone (or other glucocorticoid); Drug: Prednisone
- Control Group (Active Comparator)
  Interventions: Drug: Cyclophosphamide plus rituximab placebo (control group); Drug: Azathioprine; Drug: Methylprednisolone (or other glucocorticoid); Drug: Prednisone

INTERVENTIONS:
Drug: Rituximab plus cyclophosphamide placebo (rituximab group) — 375 mg/m^2 infusions once weekly for 4 week
  Other Names: Rituxan
  Arms: Rituximab
Drug: Cyclophosphamide plus rituximab placebo (control group) — 2 mg/kg/day orally for months 1-3
  Other Names: Cytoxan
  Arms: Control Group
Drug: Azathioprine — 2 mg/kg/day orally for months 4-6
  Other Names: imuran
  Arms: Control Group
Drug: Methylprednisolone (or other glucocorticoid) — 1 g/day intravenously for up to 3 days within 14 days prior to receiving rituximab
  Other Names: Medrol
Drug: Prednisone — During the remission induction phase, all participants will receive oral prednisone daily (1 mg/kg/day, not to exceed 80 mg/day). Prednisone tapering will be completed by the Month 6 study visit.
  Other Names: Deltasone, Liquid Pred, Meticorten, Orasone

SUMMARY:
Antineutrophil cytoplasmic antibodies (ANCA)-associated vasculitis is the most common type of small blood vessel inflammation in adults. ANCA-associated vasculitis includes Wegener's granulomatosis (WG) and microscopic polyangiitis (MPA). Rituximab is a man-made antibody used to treat certain types of cancer. The purpose of this study is to determine the effectiveness of rituximab in treating patients with WG and MPA.

Study hypothesis: Rituximab is not inferior to conventional therapy in its ability to induce disease remission by Month 6.

DETAILED DESCRIPTION:
Current conventional therapies for ANCA-associated vasculitis (AAV) are associated with high incidences of treatment failure, disease relapse, substantial toxicity, and patient morbidity and mortality. Rituximab is a monoclonal antibody used to treat non-Hodgkin's lymphoma. This study will evaluate the efficacy of rituximab with glucocorticoids in inducing disease remission in patients with severe forms of AAV (WG and MPA).

The study consists of two phases: a 6-month remission induction phase, followed by a 12-month remission maintenance phase. All participants will receive at least 1 g of pulse intravenous methylprednisolone or a dose-equivalent of another glucocorticoid preparation. Depending on the participant's condition, he or she may receive up to 3 days of intravenous methylprednisolone for a total of 3 g of methylprednisolone (or a dose-equivalent). During the remission induction phase, all participants will receive oral prednisone daily (1 mg/kg/day, not to exceed 80 mg/day). Prednisone tapering will be completed by the Month 6 study visit.

Next, participants will be randomly assigned to one of two arms. Arm 1 participants will receive rituximab (375 mg/m^2) infusions once weekly for 4 weeks and cyclophosphamide (CYC) placebo daily for 3 to 6 months. Arm 2 participants will receive rituximab placebo infusions once weekly for 4 weeks and CYC daily for 3 to 6 months. During the remission maintenance phase, participants in Arm 1 will discontinue CYC placebo and start oral azathioprine (AZA) placebo daily until Month 18. Participants in Arm 2 will discontinue CYC and start AZA daily until Month 18. Participants who fail treatment before Month 6 will be crossed over to the other treatment arm unless there are specific contraindications. Participants in either group who reach clinical remission before they complete 6 months of therapy may switch from CYC/placebo to AZA/placebo if directed by their physicians.

All participants will be followed for at least 18 months. Initially, study visits are weekly, progressing to monthly and then quarterly visits as the study proceeds. Blood collection will occur at each study visit.

ELIGIBILITY:
Inclusion Criteria:

* Weight of at least 88 pounds(40 kilograms)
* Diagnosis of Wegener's granulomatosis or microscopic polyangiitis according to the definitions of the Chapel Hill Consensus Conference
* Newly diagnosed patient of Wegener's granulomatosis or microscopic polyangiitis OR must be experiencing a disease flare characterized by: (a) active disease with a Birmingham Vasculitis Activity Score for Wegener's granulomatosis (BVAS/WG) of 3 or greater that would normally require treatment with CYC; OR (b) disease severe enough to require treatment with CYC; OR (c) must be positive for either PR3-ANCA (ANCA directed against proteinase 3) or MPO-ANCA (ANCA directed against myeloperoxidase)at the screening
* Willing to use acceptable forms of contraception for the duration of the study and for up to 1 year after stopping study medications
* Willing to report pregnancies (female participants or male participants' partners) occurring at any time during the study and for up to 1 year after stopping study medications
* Parent or guardian willing to provide informed consent, if applicable

Exclusion Criteria:

* Diagnosis of Churg-Strauss Syndrome according to the definitions of the Chapel Hill Consensus Conference
* Have limited disease that would not normally be treated with CYC
* Requires mechanical ventilation because of alveolar hemorrhage
* History of severe allergic reactions to human or chimeric monoclonal antibodies
* Active systemic infection
* Have a deep-space infection, such as osteomyelitis, septic arthritis, or pneumonia complicated by pleural cavity or lung abscess, within 6 months prior to study entry
* History of or current hepatitis B or C infection
* HIV (human immunodeficiency virus) infected
* Acute or chronic liver disease that, in the opinion of the investigator, may interfere with the study
* History of or active cancer diagnosed within the last 5 years. Individuals with squamous cell or basal cell carcinomas of the skin and individuals with cervical carcinoma in situ who have received curative surgical treatment may be eligible for this study.
* History of anti-glomerular basement membrane (anti-GBM) disease
* Other uncontrolled disease, including drug and alcohol abuse, that may interfere with the study
* Pregnancy or breastfeeding

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 197 (Actual)
Dates: Start 2005-01; Primary Completion 2008-12 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John H. Stone, MD, MPH, Study Chair — Johns Hopkins University; Ulrich Specks, MD, Study Chair — Mayo Clinic
Locations (8):
- United States (7):
  - University of Alabama, Birmingham, Alabama
  - Johns Hopkins University, Baltimore, Maryland
  - Boston University, Boston, Massachusetts
  - Mayo Clinic Foundation, Rochester, Minnesota
  - Hospital for Special Surgery, New York, New York
  - Duke University, Durham, North Carolina
  - The Cleveland Clinic, Cleveland, Ohio
- University Hospital Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Participant level data and additional relevant materials are available to the public in: 1.) the Immunology Database and Analysis Portal (ImmPort), a long-term archive of clinical and mechanistic data from DAIT-funded grants and contracts; and 2.) TrialShare, the Immune Tolerance Network (ITN) Clinical Trials Research Portal.

REFERENCES:
- [Background] Zarin DA. Participant-level data and the new frontier in trial transparency. N Engl J Med. 2013 Aug 1;369(5):468-9. doi: 10.1056/NEJMe1307268. No abstract available. PMID 23902488
- [Result] Stone JH, Merkel PA, Spiera R, Seo P, Langford CA, Hoffman GS, Kallenberg CG, St Clair EW, Turkiewicz A, Tchao NK, Webber L, Ding L, Sejismundo LP, Mieras K, Weitzenkamp D, Ikle D, Seyfert-Margolis V, Mueller M, Brunetta P, Allen NB, Fervenza FC, Geetha D, Keogh KA, Kissin EY, Monach PA, Peikert T, Stegeman C, Ytterberg SR, Specks U; RAVE-ITN Research Group. Rituximab versus cyclophosphamide for ANCA-associated vasculitis. N Engl J Med. 2010 Jul 15;363(3):221-32. doi: 10.1056/NEJMoa0909905. PMID 20647199
- [Result] Specks U, Merkel PA, Seo P, Spiera R, Langford CA, Hoffman GS, Kallenberg CG, St Clair EW, Fessler BJ, Ding L, Viviano L, Tchao NK, Phippard DJ, Asare AL, Lim N, Ikle D, Jepson B, Brunetta P, Allen NB, Fervenza FC, Geetha D, Keogh K, Kissin EY, Monach PA, Peikert T, Stegeman C, Ytterberg SR, Mueller M, Sejismundo LP, Mieras K, Stone JH; RAVE-ITN Research Group. Efficacy of remission-induction regimens for ANCA-associated vasculitis. N Engl J Med. 2013 Aug 1;369(5):417-27. doi: 10.1056/NEJMoa1213277. PMID 23902481
- [Result] Miloslavsky EM, Specks U, Merkel PA, Seo P, Spiera R, Langford CA, Hoffman GS, Kallenberg CG, St Clair EW, Tchao NK, Viviano L, Ding L, Sejismundo LP, Mieras K, Ikle D, Jepson B, Mueller M, Brunetta P, Allen NB, Fervenza FC, Geetha D, Keogh K, Kissin EY, Monach PA, Peikert T, Stegeman C, Ytterberg SR, Stone JH; Rituximab in ANCA-Associated Vasculitis-Immune Tolerance Network Research Group. Clinical outcomes of remission induction therapy for severe antineutrophil cytoplasmic antibody-associated vasculitis. Arthritis Rheum. 2013 Sep;65(9):2441-9. doi: 10.1002/art.38044. PMID 23754238
- [Result] Monach PA, Warner RL, Tomasson G, Specks U, Stone JH, Ding L, Fervenza FC, Fessler BJ, Hoffman GS, Ikle D, Kallenberg CG, Krischer J, Langford CA, Mueller M, Seo P, St Clair EW, Spiera R, Tchao N, Ytterberg SR, Johnson KJ, Merkel PA. Serum proteins reflecting inflammation, injury and repair as biomarkers of disease activity in ANCA-associated vasculitis. Ann Rheum Dis. 2013 Aug;72(8):1342-50. doi: 10.1136/annrheumdis-2012-201981. Epub 2012 Sep 12. PMID 22975753
- [Result] Nasrallah M, Pouliot Y, Hartmann B, Dunn P, Thomson E, Wiser J, Butte AJ. Reanalysis of the Rituximab in ANCA-Associated Vasculitis trial identifies granulocyte subsets as a novel early marker of successful treatment. Arthritis Res Ther. 2015 Sep 21;17(1):262. doi: 10.1186/s13075-015-0778-z. PMID 26387933
- [Result] Miloslavsky EM, Specks U, Merkel PA, Seo P, Spiera R, Langford CA, Hoffman GS, Kallenberg CG, St Clair EW, Tchao NK, Ding L, Ikle D, Villareal M, Lim N, Brunetta P, Fervenza FC, Monach PA, Stone JH; Rituximab in ANCA-Associated Vasculitis-Immune Tolerance Network Research Group. Outcomes of nonsevere relapses in antineutrophil cytoplasmic antibody-associated vasculitis treated with glucocorticoids. Arthritis Rheumatol. 2015 Jun;67(6):1629-36. doi: 10.1002/art.39104. PMID 25776953
- [Result] Miloslavsky EM, Specks U, Merkel PA, Seo P, Spiera R, Langford CA, Hoffman GS, Kallenberg CG, St Clair EW, Tchao NK, Viviano L, Ding L, Ikle D, Villarreal M, Jepson B, Brunetta P, Allen NB, Fervenza FC, Geetha D, Keogh K, Kissin EY, Monach PA, Peikert T, Stegeman C, Ytterberg SR, Stone JH; Rituximab in ANCA-Associated Vasculitis-Immune Tolerance Network Research Group. Rituximab for the treatment of relapses in antineutrophil cytoplasmic antibody-associated vasculitis. Arthritis Rheumatol. 2014 Nov;66(11):3151-9. doi: 10.1002/art.38788. PMID 25047592
- [Derived] Berti A, Hillion S, Hummel AM, Son YM, Chriti N, Peikert T, Carmona EM, Abdulahad WH, Heeringa P, Harris KM, St Clair EW, Brunetta P, Fervenza FC, Langford CA, Kallenberg CG, Merkel PA, Monach PA, Seo P, Spiera RF, Stone JH, Grandi G, Sun J, Pers JO, Specks U, Cornec D; RAVE-ITN Research Group. Circulating autoreactive proteinase 3+ B cells and tolerance checkpoints in ANCA-associated vasculitis. JCI Insight. 2021 Nov 22;6(22):e150999. doi: 10.1172/jci.insight.150999. PMID 34618687
- [Derived] Kronbichler A, Leierer J, Shin JI, Merkel PA, Spiera R, Seo P, Langford CA, Hoffman GS, Kallenberg CGM, St Clair EW, Brunetta P, Fervenza FC, Geetha D, Keogh KA, Monach PA, Ytterberg SR, Mayer G, Specks U, Stone JH; RAVE-ITN Research Group. Association of Pulmonary Hemorrhage, Positive Proteinase 3, and Urinary Red Blood Cell Casts With Venous Thromboembolism in Antineutrophil Cytoplasmic Antibody-Associated Vasculitis. Arthritis Rheumatol. 2019 Nov;71(11):1888-1893. doi: 10.1002/art.41017. Epub 2019 Sep 25. PMID 31216123
- [Derived] Wallace ZS, Miloslavsky EM, Cascino M, Unizony SH, Lu N, Hoffman GS, Kallenberg CGM, Langford CA, Merkel PA, Monach PA, Seo P, Spiera R, St Clair EW, Specks U, Brunetta P, Choi HK, Stone JH. Effect of Disease Activity, Glucocorticoid Exposure, and Rituximab on Body Composition During Induction Treatment of Antineutrophil Cytoplasmic Antibody-Associated Vasculitis. Arthritis Care Res (Hoboken). 2017 Jul;69(7):1004-1010. doi: 10.1002/acr.23099. PMID 27696762
- [Derived] Unizony S, Villarreal M, Miloslavsky EM, Lu N, Merkel PA, Spiera R, Seo P, Langford CA, Hoffman GS, Kallenberg CM, St Clair EW, Ikle D, Tchao NK, Ding L, Brunetta P, Choi HK, Monach PA, Fervenza F, Stone JH, Specks U; RAVE-ITN Research Group. Clinical outcomes of treatment of anti-neutrophil cytoplasmic antibody (ANCA)-associated vasculitis based on ANCA type. Ann Rheum Dis. 2016 Jun;75(6):1166-9. doi: 10.1136/annrheumdis-2015-208073. Epub 2015 Nov 30. PMID 26621483
- See also: National Institute of Allergy and Infectious Diseases (NIAID) website — https://www.niaid.nih.gov/
- See also: Division of Allergy, Immunology, and Transplantation (DAIT) website — https://www.niaid.nih.gov/about/dait
- See also: Immune Tolerance Network website — http://www.immunetolerance.org
- See also: Genentech website — https://www.gene.com/
- Available data/document: Individual Participant Data Set: SDY91 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY91 — ImmPort study identifier is SDY91.
- Available data/document: Study summary, -design, -adverse event(s), -summary of participant assessments, -interventions, -medications, -demographics, -lab tests, -mechanistic assays, -files et al.: SDY91 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY91 — ImmPort study identifier is SDY91.
- Available data/document: Individual Participant Data Set: ITN021AI — https://www.itntrialshare.org/project/home/begin.view? — TrialShare study ID is ITN021AI.
- Available data/document: Study overview, -data and reports, -participant list, -manuscripts and abstracts, -availability of biospecimens.: ITN021AI — https://www.itntrialshare.org/project/home/begin.view? — TrialShare study ID is ITN021AI.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eight centers in the United States and one center in the Netherlands (Groningen) enrolled 197 Antineutrophil cytoplasmic antibodies (ANCA)-positive patients with either Wegener's granulomatosis or microscopic polyangiitis between December 30, 2004 and June 30, 2008.
Pre-assignment Details: At a screening visit, participants underwent procedures to establish inclusion/exclusion criteria and then sign the informed consent form.
Groups:
- Rituximab: Participants received intravenous rituximab (Rituxan, Genentech) (at a dose of 375 mg per square meter of body-surface area once weekly for 4 weeks) plus daily placebo-cyclophosphamide. Refer to section titled "Detailed Description" for additional treatment information.
- Control Group: Participants received placebo-rituximab infusions plus daily cyclophosphamide (2 mg per kilogram of body weight, adjusted for renal insufficiency). Refer to section titled "Detailed Description" for additional treatment information.
Period: Overall Study
Arm/Group | Rituximab | Control Group
Started | 99 | 98
Completed | 90 (Number of participants who completed 18 months post-randomization) | 88 (Number of participants who completed 18 months post-randomization)
Not Completed | 9 | 10
Not completed — Adverse Event | 3 | 1
Not completed — Death | 2 | 2
Not completed — Withdrawal by Subject | 2 | 6
Not completed — Physician Decision | 1 | 1
Not completed — To have renal transplant | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rituximab | Control Group | Total
Number analyzed (Participants) | 99 | 98 | 197
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3 | 3 | 6
  Between 18 and 65 years | 60 | 76 | 136
  >=65 years | 36 | 19 | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.0 (16.8) | 51.5 (14.1) | 52.8 (15.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 45 | 97
  Male | 47 | 53 | 100
Region of Enrollment [Number; unit: participants]
  United States | 91 | 90 | 181
  Netherlands | 8 | 8 | 16
BVAS/WG [Mean (Standard Deviation); unit: score units] — The Birmingham Vasculitis Activity Score for Wegener's Granulomatosis (WG) is a validated disease activity index. The BVAS/WG is designed to document new or worsening clinically active vasculitis and consists of a set of items divided into nine organ based systems. BVAS/WG scores range from 0 to 63, with higher scores indicating more active disease. In this study, the primary end point was a BVAS/WG score of 0 and successful completion of the prednisone taper at 6 months.
  score units | 8.1 (2.8) | 8.0 (3.4) | 8.0 (3.1)
VDI [Mean (Standard Deviation); unit: score units] — Vasculitis Damage Index. The VDI is a validated measure for damage assessment in vasculitis. The index comprises 64 items of damage (divided into 11 organ based systems) representative of damage incurred to patients with systemic vasculitis. Scores for this index range from 0 to 64, with higher scores indicating more severe damage.
  score units | 1.4 (1.8) | 1.0 (1.4) | 1.2 (1.7)

OUTCOME MEASURES:

1. Primary Outcome: Disease Remission
Description: A Birmingham Vasculitis Activity Score for Wegener's Granulomatosis (BVAS/WG) score of 0 with prednisone taper successfully completed at six months. The BVAS/WG is a validated disease activity index. The BVAS/WG is designed to document new or worsening clinically active vasculitis and consists of a set of items divided into nine organ based systems. BVAS/WG scores range from 0 to 63, with higher scores indicating more active disease.
Time Frame: 6 months post-randomization
Population: Intent-to-treat (ITT) sample with worst case imputation
Measure: Number; unit: Participants
Arm/Group | Rituximab | Control Group
Number analyzed (Participants) | 99 | 98
Participants | 63 | 52
Statistical Analysis 1: Comparison: Rituximab vs Control Group; In calculating the sample size, we assumed that the percentage of patients in both treatment groups would achieve disease remission off prednisone by 6 months was 70%. We specified a non-inferiority margin of -20% on the difference in remission rates (rituximab rate minus cyclophosphamide rate) and a one-sided 0.025 level test. Assuming a 10% dropout rate, RAVE required 100 patients in each arm to have 83% power to conclude non-inferiority; Test type: Non-Inferiority or Equivalence — non-inferiority margin of -20%; p < 0.001, 95.1% CI of difference — P-value is adjusted for interim analysis using a Lan-DeMets alpha spending function with an O'Brien-Fleming boundary, allocating 0.003 alpha to the interim analysis and 0.049 alpha to the final analysis; Calculate 95.1% CI around the difference in success rates between arms. Lower bound above non-inferiority margin of -20% indicates non-inferiority; Difference between group success rates = 10.6, 95.1% CI [-3.2 to 24.3]

2. Secondary Outcome: Rate of Selected Adverse Events Experienced by Participants Receiving Rituximab Versus Those Receiving Conventional Therapy
Description: The adverse event rate for the following events considered related to vasculitis: Death; Grade 2 or higher leukopenia or thrombocytopenia; Grade 3 or higher infections; Hemorrhagic cystitis (grade 2 or lower needs confirmation by cytoscopy); Malignancy; Venous thromboembolic event (deep venous thrombosis or pulmonary embolism); Hospitalization resulting either from the disease or from a complication due to study treatment; Infusion reactions (within 24 hours of infusion) that result in the cessation of further infusions (including cytokine release allergic reaction); Cerebrovascular accident
Time Frame: Through common close-out (defined as 18 months after the last participant is enrolled in the trial)
Population: Safety Sample
Measure: Number; unit: participants
Arm/Group | Rituximab | Control Group
Number analyzed (Participants) | 99 | 98
participants
  Death | 2 | 2
  Grade 2 or Higher Leukopenia | 7 | 23
  Grade 2 or Higher Thrombocytopenia | 4 | 1
  Grade 3 or Higher Infections | 18 | 16
  Hemorrhagic Cystitis (Grade 2 or Lower) | 2 | 1
  Malignancy | 5 | 2
  Venous Thromboembolic Event | 6 | 8
  Hospitalization Resulting from the Disease | 16 | 7
  Cerebrovascular Accident (CVA) | 1 | 1
  Infusion Reactions Leading to Infusion Disc. | 1 | 0
Statistical Analysis 1: Comparison: Rituximab vs Control Group; Participant-months are defined as duration in months from the first study drug dosing date to the last date of the participant in the protocol. The rate of selected AEs is defined as the total number of selected AEs divided by total participant-months, and indicates the number of events per participant per month on average. Participants are grouped according to their originally received treatment; Test type: Superiority or Other; p = 0.927, Poisson regression model — P-value is from the Poisson regression model adjusting for clinical study site and ANCA type. The natural logarithm of participant-months is used as an offset in this model

3. Secondary Outcome: Percentage of Participants Who Have a BVAS/WG Score of 0 and Have Successfully Completed the Glucocorticoid Taper by 6 Months Post-randomization
Description: The 2-sided 95% CI of the percentage of participants who have a Birmingham Vasculitis Activity Score for Wegener's Granulomatosis (BVAS/WG)[1] of 0 and have successfully completed the glucocorticoid taper by 6 months post-randomization and the 2-sided 95% CI of the difference between two arms for assessing the superiority of rituximab to control
  [1] The BVAS/WG is a disease activity index designed to document new or worsening clinically active vasculitis consisting of items divided into 9 organ based systems. BVAS/WG scores range from 0 to 63, with higher scores indicating more active disease
Time Frame: 6 months post-randomization
Population: Safety Sample
Measure: Number; unit: participants
Arm/Group | Rituximab | Control Group
Number analyzed (Participants) | 99 | 98
participants | 62 | 51
Statistical Analysis 1: Comparison: Rituximab vs Control Group; The p-value is from a chi-square test; Test type: Superiority or Other; p = 0.133, Chi-squared; At 6 months, the confidence interval is 95.1%; 95.1% Confidence Interval of Difference = 10.6, 95.1% CI 2-sided [-3.2 to 24.4]

4. Secondary Outcome: The Duration of Complete Remission (BVAS=0, Off Glucocorticoids), the Time to Limited and/or Severe Flare After Remission in the Two Treatment Groups
Description: Duration of complete remission is defined as a Birmingham Vasculitis Activity Score for Wegener's Granulomatosis (BVAS/WG)[1] of 0 and a completing taper of Prednisone to the first flare, BVAS/WG score of greater than 0, or an increase in Prednisone dosing.
  [1] The BVAS/WG is a disease activity index designed to document new or worsening clinically active vasculitis consisting of items divided into 9 organ based systems. BVAS/WG scores range from 0 to 63, with higher scores indicating more active disease
Time Frame: 18 months post-randomization
Population: Intent-to-treat
Measure: Number (95% Confidence Interval); unit: Days
Arm/Group | Rituximab | Control Group
Number analyzed (Participants) | 99 | 98
Days
  25% Quartile (95%CI) | 243 [172 to NA] — Some survival parameters are not estimable when there are small numbers of events | 230 [145 to NA] — Some survival parameters are not estimable when there are small numbers of events
  50% Quartile (95%CI) | NA [NA to NA] — Some survival parameters are not estimable when there are small numbers of events | NA [NA to NA] — Some survival parameters are not estimable when there are small numbers of events
  75% Quartile (95%CI) | NA [NA to NA] — Some survival parameters are not estimable when there are small numbers of events | NA [NA to NA] — Some survival parameters are not estimable when there are small numbers of events
Statistical Analysis 1: Comparison: Rituximab vs Control Group; Participants are censored at the time of crossover, open label rituximab, or best medical judgement, if applicable. If a participant has no flare after complete remission prior to their Month 18 visit, the duration is censored at the date of the Month 18 Visit; Test type: Superiority or Other; p = 0.761, Log Rank — The log-rank test assesses the difference between the two treatment arms in the flaring pattern after complete remission; The log-rank test assesses the difference between the two treatment arms in the flaring pattern after complete remission; Cox Proportional Hazard = 0.9, 95% CI 2-sided [0.5 to 1.7]

5. Secondary Outcome: The Duration of Remission (BVAS=0), the Time to Limited and/or Severe Flare After Remission in the Two Treatment Groups
Description: Duration of remission is defined as a Birmingham Vasculitis Activity Score for Wegener's Granulomatosis (BVAS/WG)[1] of 0 and a completing taper of glucocorticoid by 6 months post-randomization to the first flare, BVAS/WG score of greater than 0, or an increase in Prednisone dosing.
Time Frame: 18 months post-randomization
Population: Intent-to-treat
Measure: Number (95% Confidence Interval); unit: Days
Arm/Group | Rituximab | Control Group
Number analyzed (Participants) | 99 | 98
Days
  25% Quartile (95%CI) | 246 [152 to 335] | 168 [141 to 300]
  50% Quartile (95%CI) | NA [403 to NA] — Some survival parameters are not estimable when there are small numbers of events | NA [353 to NA] — Some survival parameters are not estimable when there are small numbers of events
  75% Quartile (95%CI) | NA [NA to NA] — Some survival parameters are not estimable when there are small numbers of events | NA [NA to NA] — Some survival parameters are not estimable when there are small numbers of events
Statistical Analysis 1: Comparison: Rituximab vs Control Group; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.861, Log Rank; The log-rank test assesses the difference between the two treatment arms in the flaring pattern after remission; Cox Proportional Hazard = 0.9, 95% CI 2-sided [0.6 to 1.5]

6. Secondary Outcome: Time to Remission (BVAS=0) From the Visit 1 Baseline Visit in the Two Treatment Groups
Description: Time to complete remission is defined as the number of days from baseline visit (Visit 1) to a Birmingham Vasculitis Activity Score for Wegener's Granulomatosis (BVAS/WG)[1] of 0.
  [1] The BVAS/WG is a disease activity index designed to document new or worsening clinically active vasculitis consisting of items divided into 9 organ based systems. BVAS/WG scores range from 0 to 63, with higher scores indicating more active disease
Time Frame: 18 months post-randomization
Population: Intent-to-treat
Measure: Number (95% Confidence Interval); unit: Days
Arm/Group | Rituximab | Control Group
Number analyzed (Participants) | 99 | 98
Days
  25% Quartile (95%CI) | 30 [29 to 34] | 29 [NA to NA] — Confidence limits not estimable due to no variability around quartile
  50% Quartile (95%CI) | 57 [41 to 63] | 43 [30 to 58]
  75% Quartile (95%CI) | 119 [69 to 123] | 112 [61 to 120]
Statistical Analysis 1: Comparison: Rituximab vs Control Group; Test type: Superiority or Other; p = 0.497, Log Rank; The log-rank test assesses the difference between the two treatment arms in the pattern of achieving remission; Cox Proportional Hazard = 1.0, 95% CI 2-sided [0.7 to 1.3] — The hazard ratio and confidence interval are based on a Cox proportional hazard model comparing rituximab to the control group, adjusting for clinical study site, ANCA type, and glucocorticoid use prior to baseline

7. Secondary Outcome: Time to Complete Remission (BVAS=0, Off Glucocorticoids) From the Visit 1 Baseline Visit in the Two Treatment Groups
Description: Time to complete remission is defined as the number of days from baseline visit (Visit 1) to a Birmingham Vasculitis Activity Score for Wegener's Granulomatosis (BVAS/WG)[1] of 0 and completing taper of glucocorticoid by 6 months post-randomization.
  [1] The BVAS/WG is a disease activity index designed to document new or worsening clinically active vasculitis consisting of items divided into 9 organ based systems. BVAS/WG scores range from 0 to 63, with higher scores indicating more active disease
Time Frame: 18 months post-randomization
Population: Intent-to-treat
Measure: Number (95% Confidence Interval); unit: Days
Arm/Group | Rituximab | Control Group
Number analyzed (Participants) | 99 | 98
Days
  25% Quartile (95%CI) | 176 [173 to 177] | 177 [175 to 178]
  50% Quartile (95%CI) | 180 [178 to 182] | 183 [180 to 187]
  75% Quartile (95%CI) | 189 [183 to 253] | 266 [190 to 287]
Statistical Analysis 1: Comparison: Rituximab vs Control Group; Test type: Superiority or Other; p = 0.147, Log Rank; The log-rank test assesses the difference between the two treatment arms in the pattern of achieving complete remission; Cox Proportional Hazard = 1.3, 95% CI 2-sided [0.9 to 1.8] — [estimate comment as in outcome 6, analysis 1]

8. Post Hoc Outcome: Number of Subjects Experiencing Serious Adverse Events
Description: Number of subjects according to originally received treatment that experienced a serious adverse event through 18 months post-randomization or prior to being censored from analyses due to crossover, switching to open-label treatment, or best medical judgment for censor. Events are categorized by coded system organ classes (SOC). Within each SOC, a participant was counted once if the participant reported one or more events coded to that SOC.
Time Frame: Randomization to censor at Crossover, Open-label or Best Medical Judgment (up to 18 months post-randomization)
Population: Intent-to-treat
Measure: Number; unit: participants
Arm/Group | Rituximab | Control Group
Number analyzed (Participants) | 99 | 98
participants
  # Participants with at least one SAE | 42 | 37
  Blood and Lymphatic System Disorders | 4 | 5
  Cardiac Disorders | 2 | 2
  Eye Disorders | 1 | 1
  Gastrointestinal Disorders | 4 | 1
  General Disorders and Administration Site | 5 | 3
  Immune System Disorders | 2 | 2
  Infections and Infestations | 12 | 12
  Injury, Poisoning, and Procedural Complications | 2 | 0
  Investigations | 2 | 0
  Metabolism and Nutrition Disorders | 2 | 2
  Musculoskeletal and Connective Tissue Disorders | 2 | 3
  Neoplasms Benign, Malignant, and Unspecified | 1 | 2
  Nervous System Disorders | 1 | 0
  Pregnancy, Puerperium, and Perinatal Conditions | 1 | 0
  Psychiatric Disorders | 1 | 1
  Renal and Urinary Disorders | 4 | 3
  Respiratory, Thoracic, and Mediastinal Disorders | 8 | 8
  Vascular Disorders | 1 | 7
Statistical Analysis 1: Comparison: Rituximab vs Control Group; Proportions of subjects experiencing a serious adverse event through 18 months and prior to censoring for open-label, crossover, or best medical judgment according to originally assigned treatment arm were compared using a two-sided Chi-squared test; Test type: Superiority or Other; p = 0.504, Chi-squared

ADVERSE EVENTS:
Time Frame: From randomization through common close out (defined as 18 months after the last participant is enrolled in the trial)
Description: Adverse events reported include both disease and non-disease related events by originally assigned treatment. No participants are censored from these results. NCI-CTCAE version 3.0 (published June 10, 2003) was used to grade severity.
Arm/Group | Rituximab | Control Group
Serious Adverse Events (participants affected / at risk) | 60/99 | 47/98
Other Adverse Events (participants affected / at risk) | 97/99 | 97/98
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rituximab (N=99) | Control Group (N=98)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 4 (6)
Autoimmune thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Leukopenia (Blood and lymphatic system disorders) | 3 (5) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 0 (0)
Atrial tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Sudden hearing loss (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Keratitis (Eye disorders) | 1 (1) | 0 (0)
Ulcerative keratitis (Eye disorders) | 0 (0) | 1 (1)
Colitis ischaemic (Gastrointestinal disorders) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Impaired gastric emptying (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 2 (2)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Adverse drug reaction (General disorders) | 1 (1) | 1 (1)
Asthenia (General disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 1 (1)
Chills (General disorders) | 0 (0) | 2 (2)
Multi-organ failure (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Anti-neutrophil cytoplasmic antibody positive vasculitis (Immune system disorders) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 2 (2)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Abdominal abscess (Infections and infestations) | 1 (1) | 0 (0)
Abscess limb (Infections and infestations) | 1 (1) | 0 (0)
Acute sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis orbital (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis staphylococcal (Infections and infestations) | 1 (1) | 0 (0)
Central line infection (Infections and infestations) | 0 (0) | 1 (1)
Clostridial infection (Infections and infestations) | 1 (2) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0)
Escherichia infection (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 1 (1)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Lobar pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0)
Periorbital cellulitis (Infections and infestations) | 0 (0) | 1 (2)
Pneumocystis jiroveci pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 8 (10) | 10 (11)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1)
Post streptococcal glomerulonephritis (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 1 (1)
C-reactive protein increased (Investigations) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypovolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Bone disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (6)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0)
Acute prerenal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Bladder disorder (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 1 (1)
Renal failure (Renal and urinary disorders) | 4 (4) | 2 (2)
Renal failure acute (Renal and urinary disorders) | 2 (2) | 3 (3)
Renal failure chronic (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Endometriosis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Laryngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (3)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Wegener's granulomatosis (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 4 (5)
Aortic dissection (Vascular disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 8 (8)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rituximab (N=99) | Control Group (N=98)
Anaemia (Blood and lymphatic system disorders) | 22 (28) | 18 (23)
Leukopenia (Blood and lymphatic system disorders) | 13 (30) | 39 (80)
Thrombocytopenia (Blood and lymphatic system disorders) | 9 (13) | 5 (6)
Ear pain (Ear and labyrinth disorders) | 7 (8) | 5 (5)
Cushingoid (Endocrine disorders) | 5 (6) | 6 (6)
Vision blurred (Eye disorders) | 4 (4) | 7 (7)
Diarrhoea (Gastrointestinal disorders) | 27 (35) | 20 (25)
Dyspepsia (Gastrointestinal disorders) | 7 (7) | 8 (8)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 10 (10) | 6 (6)
Nausea (Gastrointestinal disorders) | 25 (28) | 31 (41)
Vomiting (Gastrointestinal disorders) | 8 (12) | 13 (18)
Chest discomfort (General disorders) | 6 (7) | 4 (4)
Chest pain (General disorders) | 6 (6) | 4 (4)
Chills (General disorders) | 6 (7) | 5 (5)
Fatigue (General disorders) | 26 (32) | 30 (42)
Oedema peripheral (General disorders) | 22 (26) | 14 (19)
Pyrexia (General disorders) | 10 (12) | 17 (25)
Bronchitis (Infections and infestations) | 7 (11) | 8 (11)
Herpes zoster (Infections and infestations) | 9 (10) | 8 (8)
Influenza (Infections and infestations) | 5 (6) | 5 (5)
Nasopharyngitis (Infections and infestations) | 11 (18) | 14 (22)
Sinusitis (Infections and infestations) | 16 (28) | 17 (29)
Upper respiratory tract infection (Infections and infestations) | 29 (43) | 24 (40)
Urinary tract infection (Infections and infestations) | 18 (24) | 7 (10)
Viral upper respiratory tract infection (Infections and infestations) | 7 (8) | 4 (4)
Alanine aminotransferase increased (Investigations) | 15 (23) | 22 (30)
Aspartate aminotransferase increased (Investigations) | 11 (14) | 16 (21)
Blood creatinine increased (Investigations) | 8 (10) | 10 (12)
C-reactive protein increased (Investigations) | 8 (10) | 9 (11)
Haematocrit decreased (Investigations) | 8 (8) | 16 (19)
Haemoglobin decreased (Investigations) | 6 (7) | 7 (8)
Red blood cell sedimentation rate increased (Investigations) | 5 (9) | 12 (14)
Weight increased (Investigations) | 6 (8) | 8 (8)
White blood cell count decreased (Investigations) | 6 (9) | 21 (43)
Hyperglycaemia (Metabolism and nutrition disorders) | 12 (15) | 11 (11)
Hyperkalaemia (Metabolism and nutrition disorders) | 8 (19) | 5 (6)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (4) | 7 (9)
Arthralgia (Musculoskeletal and connective tissue disorders) | 34 (42) | 24 (34)
Back pain (Musculoskeletal and connective tissue disorders) | 13 (13) | 10 (10)
Joint swelling (Musculoskeletal and connective tissue disorders) | 8 (9) | 3 (3)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 20 (26) | 21 (23)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 6 (7) | 4 (5)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 11 (11) | 4 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (6) | 8 (8)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 13 (17) | 10 (10)
Dizziness (Nervous system disorders) | 14 (17) | 12 (16)
Dysgeusia (Nervous system disorders) | 6 (7) | 6 (6)
Headache (Nervous system disorders) | 28 (31) | 25 (41)
Hypoaesthesia (Nervous system disorders) | 9 (10) | 8 (9)
Paraesthesia (Nervous system disorders) | 4 (7) | 7 (9)
Tremor (Nervous system disorders) | 10 (15) | 6 (6)
Depression (Psychiatric disorders) | 7 (7) | 6 (6)
Insomnia (Psychiatric disorders) | 18 (20) | 14 (15)
Haematuria (Renal and urinary disorders) | 6 (8) | 14 (16)
Cough (Respiratory, thoracic and mediastinal disorders) | 32 (40) | 24 (31)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 10 (12) | 5 (7)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 16 (18) | 15 (19)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 18 (26) | 15 (23)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 8 (10) | 7 (8)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 13 (13) | 8 (9)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 11 (14) | 3 (4)
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 5 (7) | 6 (8)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 7 (11)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 5 (5)
Acne (Skin and subcutaneous tissue disorders) | 7 (9) | 5 (5)
Alopecia (Skin and subcutaneous tissue disorders) | 11 (13) | 21 (21)
Rash (Skin and subcutaneous tissue disorders) | 14 (19) | 23 (28)
Flushing (Vascular disorders) | 6 (11) | 7 (8)
Hypertension (Vascular disorders) | 14 (18) | 10 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No